CLINICAL TRIAL: NCT04694248
Title: Anticoagulant Plus Antiplatelet Therapy Following Iliac Vein Stenting
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Collaborators: Zhejiang University (Other); Ningbo No.2 Hospital (Other); Taizhou Hospital of Zhejiang Province affiliated to Wenzhou Medical University (Other); The Central Hospital of Lishui City (Other); Taizhou Enze Medical Center Group (Other); Taizhou First People's Hospital (Other); Boston Scientific Corporation (Industry)
Responsible Party: Principal Investigator, Hongkun Zhang, MD, Chief of Department of Vascular Surgery, First Affiliated Hospital of Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT20200040C
Record Dates: First submitted 2021-01-01; First posted 2021-01-05 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Deep Vein Thrombosis; Iliac Vein Thrombosis; Iliac Vein Obstruction; Iliac Vein Stenosis; Iliac Vein Compression Syndrome
Keywords: acute proximal deep vein thrombosis; iliac vein stenting
MeSH Terms: conditions — Venous Thrombosis; May-Thurner Syndrome | interventions — Rivaroxaban; Anticoagulants; Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Anticoagulant plus antiplatelet therapy (Experimental): For anticoagulant, it is rivaroxaban 20mg once a day for 6 months. For antiplatelet therapy, it is aspirin 100mg once a day indefinitely.
  Interventions: Drug: Rivaroxaban; Drug: Aspirin

INTERVENTIONS:
Drug: Rivaroxaban — For anticoagulant, it is rivaroxaban 20mg once a day for 6 months.
  Other Names: Anticoagulant
Drug: Aspirin — For antiplatelet therapy, it is aspirin 100mg once a day indefinitely.
  Other Names: Antiplatelet

SUMMARY:
To evaluate the efficacy and safety of combination of anticoagulant and antiplatelet therapy on the patency of iliac vein at 12-month post stenting in patients with acute proximal DVT and ipsilateral iliac vein stenosis who received percutaneous mechanic thrombectomy and iliac vein stenting.

DETAILED DESCRIPTION:
This study is a single-arm, prospective, open-label, multicenter study conducted in the Zhejiang Province, China. Randomized controlled trial is not an optimum option at this stage given the lack of high-quality data in terms of this hypothesis. Eligible subjects will include men and women with age of 18 years or older, who have a confirmed diagnosis of acute proximal DVT with ipsilateral iliac vein stenosis. A total of 172 subjects will be enrolled. The inclusion criteria and exclusion criteria are pre-defined. Subjects meeting all inclusion and no exclusion criteria will be eligible for enrollment. All subjects will receive the combination of anticoagulant and antiplatelet therapy after implanted with iliac vein stent. For anticoagulant, it is rivaroxaban 20mg once a day for 6 months. For antiplatelet therapy, it is aspirin 100mg once a day indefinitely.The duration of study participation for each subject is 12 months. Each subject will be followed at 3 months, 6 months and 12 months post-procedure. Efficacy endpoints and safety endpoints will be documented during the follow-up. After completing the follow-up, data will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

IC1. Subjects who were diagnosed with deep venous thrombus (DVT) with ipsilateral iliac venous stenosis (>50%). The ipsilateral iliac venous stenosis can be caused either by iliac vein compression (i.e. Cockett syndrome) or residue iliac venous thrombus after percutaneous mechanic thrombectomy.

IC2. Subjects who accepted percutaneous mechanic thrombectomy (PMT) to decrease the burden of thrombus, with or without catheter directed thrombolysis (CDT).

IC3. Subjects who accepted iliac venous stent(s) implantation during the perioperative period of PMT or CDT (≤30 days post PMT or CDT) .

Exclusion Criteria:

EC1. Subject has chronic DVT or the onset of DVT is longer than 3 weeks, or chronic DVT.

EC2. Subject has isolated distal DVT, which does not affect ipsilateral femoral or iliac vein.

EC3. Subject has glomerular filtration rate < 60ml/min. EC4. Subject has ipsilateral varicose vein or suffers from ipsilateral venous insufficiency prior to the DVT. The manifestations of venous insufficiency include skin pigmentation, edema, lipodermatosclerosis and venous ulcer.

EC5. Subject has acute arterial embolism on either side or suffers from known moderate or greater stenosis at abdominal aorta, ipsilateral iliac artery and ipsilateral lower extremity artery.

EC6. Subject has known aneurysm(s) or current limiting dissection at abdominal aorta, ipsilateral iliac artery and ipsilateral lower extremity artery.

EC7. Subject has contraindication to antiplatelet drugs or anticoagulants. EC8. Subject has systemic disease(s) that cannot be treated by current medicine.

EC9. Subject has been taking anticoagulants or antiplatelet drugs for other diseases prior to the DVT.

EC10. Subject less than 18 years old or rejected to join this study. EC11. Subject has myocardial infarction during the past 6 months. EC12. EC12. Subject who is at high bleeding risk*.

* Subject who has at least one of the below conditions will be considered at high bleeding risk: Primary history of intracerebral haemorrhage or ischemic stroke, history of other intracranial pathology, recent gastrointestinal bleeding or anaemia due to possible gastrointestinal blood loss, other gastrointestinal pathology associated with increased bleeding risk, liver failure, bleeding diathesis or coagulopathy, extreme old age or frailty, or renal failure requiring dialysis or with eGFR <15ml/min/1.73 m2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Estimated)
Dates: Start 2021-11-03 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Primary Effectiveness Endpoints | 12-month follow-up
  The primary patency at 12-month follow-up evaluated by DUS
Primary Safety Endpoints | 12-month follow-up
  The rate of major bleeding events (BARC type 5 or type 3) based on BARC definitions at 12-month follow-up.

SECONDARY OUTCOMES:
Patency | 3-month and 6-month follow-up
  The primary patency at 3-month and 6-month follow-up
The rate of bleeding events | 3-month, 6-month and 12-month follow-up
  The rate of bleeding events based on BARC definitions at 3-month, 6-month and 12-month follow-up
The rate and severity of post-thrombotic syndrome | 3-month, 6-month and 12-month follow-up
  The rate and severity of post-thrombotic syndrome (Villalta score) at 3-month, 6-month and 12-month follow-up
The recurrence rate of deep venous thrombosis | 3-month, 6-month and 12-month follow-up
  The recurrence rate of deep venous thrombosis evaluated by DUS at 3-month, 6-month and 12-month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Hongkun Zhang, M.D., Principal Investigator — First Affiliated Hospital of Zhejiang University
Locations (1):
- The First Affliated Hospital, Zhejiang University, School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Deitelzweig SB, Johnson BH, Lin J, Schulman KL. Prevalence of clinical venous thromboembolism in the USA: current trends and future projections. Am J Hematol. 2011 Feb;86(2):217-20. doi: 10.1002/ajh.21917. PMID 21264912
- [Background] Haig Y, Enden T, Grotta O, Klow NE, Slagsvold CE, Ghanima W, Sandvik L, Hafsahl G, Holme PA, Holmen LO, Njaaastad AM, Sandbaek G, Sandset PM; CaVenT Study Group. Post-thrombotic syndrome after catheter-directed thrombolysis for deep vein thrombosis (CaVenT): 5-year follow-up results of an open-label, randomised controlled trial. Lancet Haematol. 2016 Feb;3(2):e64-71. doi: 10.1016/S2352-3026(15)00248-3. Epub 2016 Jan 6. PMID 26853645
- [Background] Garcia MJ, Lookstein R, Malhotra R, Amin A, Blitz LR, Leung DA, Simoni EJ, Soukas PA. Endovascular Management of Deep Vein Thrombosis with Rheolytic Thrombectomy: Final Report of the Prospective Multicenter PEARL (Peripheral Use of AngioJet Rheolytic Thrombectomy with a Variety of Catheter Lengths) Registry. J Vasc Interv Radiol. 2015 Jun;26(6):777-85; quiz 786. doi: 10.1016/j.jvir.2015.01.036. Epub 2015 Mar 29. PMID 25824314
- [Background] Comerota AJ, Kearon C, Gu CS, Julian JA, Goldhaber SZ, Kahn SR, Jaff MR, Razavi MK, Kindzelski AL, Bashir R, Patel P, Sharafuddin M, Sichlau MJ, Saad WE, Assi Z, Hofmann LV, Kennedy M, Vedantham S; ATTRACT Trial Investigators. Endovascular Thrombus Removal for Acute Iliofemoral Deep Vein Thrombosis. Circulation. 2019 Feb 26;139(9):1162-1173. doi: 10.1161/CIRCULATIONAHA.118.037425. PMID 30586751
- [Background] Razavi MK, Jaff MR, Miller LE. Safety and Effectiveness of Stent Placement for Iliofemoral Venous Outflow Obstruction: Systematic Review and Meta-Analysis. Circ Cardiovasc Interv. 2015 Oct;8(10):e002772. doi: 10.1161/CIRCINTERVENTIONS.115.002772. PMID 26438686
- [Background] Rizvi SA, Ascher E, Hingorani A, Marks N. Stent patency in patients with advanced chronic venous disease and nonthrombotic iliac vein lesions. J Vasc Surg Venous Lymphat Disord. 2018 Jul;6(4):457-463. doi: 10.1016/j.jvsv.2018.02.004. PMID 29909853
- [Background] Milinis K, Thapar A, Shalhoub J, Davies AH. Antithrombotic Therapy Following Venous Stenting: International Delphi Consensus. Eur J Vasc Endovasc Surg. 2018 Apr;55(4):537-544. doi: 10.1016/j.ejvs.2018.01.007. Epub 2018 Feb 12. PMID 29449145
- [Background] Gurbel PA, Fox KAA, Tantry US, Ten Cate H, Weitz JI. Combination Antiplatelet and Oral Anticoagulant Therapy in Patients With Coronary and Peripheral Artery Disease. Circulation. 2019 Apr 30;139(18):2170-2185. doi: 10.1161/CIRCULATIONAHA.118.033580. PMID 31034291
- [Background] Langwieser N, Bernlochner I, Wustrow I, Dirschinger RJ, Jaitner J, Dommasch M, Bradaric C, Laugwitz KL, Ibrahim T. Combination of factor Xa inhibition and antiplatelet therapy after stenting in patients with iliofemoral post-thrombotic venous obstruction. Phlebology. 2016 Jul;31(6):430-7. doi: 10.1177/0268355515596289. Epub 2015 Jul 15. PMID 26183668
- [Background] Endo M, Jahangiri Y, Horikawa M, Kaufman JA, Schenning RC, Kolbeck KJ, Barton RE, Ohuchi Y, Liang KW, Farsad K. Antiplatelet Therapy is Associated with Stent Patency After Iliocaval Venous Stenting. Cardiovasc Intervent Radiol. 2018 Nov;41(11):1691-1698. doi: 10.1007/s00270-018-2062-5. Epub 2018 Aug 17. PMID 30120531